CLINICAL TRIAL: NCT00423605
Title: A Long-Term, Open-Label, Safety and Efficacy Study of Xyrem® (Sodium Oxybate) in Subjects With Fibromyalgia.
Brief Title: Safety and Efficacy Study of Xyrem® (Sodium Oxybate) in Subjects With Fibromyalgia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-010
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2011-10-20 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Fibromyalgia
Keywords: FMS; Fibro; Pain; Body Pain; Tenderness; Joint pain; Stiffness; Muscular Pain
MeSH Terms: conditions — Fibromyalgia; Pain; Arthralgia; Myalgia | interventions — Sodium Oxybate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Xyrem®

INTERVENTIONS:
Drug: Xyrem® — flexible dosing

SUMMARY:
The objective of this trial is to evaluate the safety and efficacy of Xyrem® in long term use.

DETAILED DESCRIPTION:
The trial is an open-label safety and efficacy study of subjects with fibromyalgia who completed either study 06-008 or 06-009. Total duration is up to 40 weeks of trial participation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has qualified for and completed either study 06-009 (NCT00423813) or 06-008 (NCT00371137).
* Subject is able, in the opinion of the investigator, to take Xyrem® for approximately 9-1/2 months.

Exclusion Criteria:

* Subject terminated early from either study 06-009 or 06-008.
* Subject experienced any serious adverse event related to study drug in either study 06-009 or 06-008.
* Subject, in the opinion of the investigator, experienced an adverse event in 06-009 or 06-008 that may prevent him/her from safely participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2006-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (91):
- United States (66):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Suncoast Internal Medicine Consultants, Auburn, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Orange County Clinical Trials, Anaheim, California
  - Northern California Research, Carmichael, California
  - Med Investigations Inc., Fair Oaks, California
  - Nerve Pro Research, Irvine, California
  - Arroyo Medical Group, Inc., Pismo Beach, California
  - AppleMed Research, Miami, Florida
  - Compass Research, Orlando, Florida
  - Sunrise Medical Research, Plantation, Florida
  - Clinical Research Group of St. Petersburg, Inc, St. Petersburg, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Center for Arthiritis and Rheumatism, Vero Beach, Florida
  - Florida Medical Clinic, P.A., Zephyhills, Florida
  - Drug Studies America, Marietta, Georgia
  - Coeur d' Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Fibromyalgia Treatment Centers of America, Chicago, Illinois
  - Deerpath Physcians Group, Gurnee, Illinois
  - Balanced Health Research Center, Peoria, Illinois
  - Graves - Gilbert Clinic, Bowling Green, Kentucky
  - Center for Arthiritis & Osteoporosis, Elizabethtown, Kentucky
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Louisiana Sleep Foundation, Baton Rouge, Louisiana
  - Capital Clinical Rsearch Asociates, Rockville, Maryland
  - FutureCare Studies, Springfield, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Professional Clinical Research, Inc. at Crystal Lake Health Center, Benzonia, Michigan
  - Professional Clinical Research, Cadillac, Michigan
  - Professional Clinical Research at Crystal Lake Health Center, Interlocken, Michigan
  - PCM Medical Services, Lansing, Michigan
  - Clinvest, Springfield, Missouri
  - School of Osteopathic Medicine, Cherry Hill, New Jersey
  - Anderson & Collins Clinical Research, Inc., Edison, New Jersey
  - Upstate Clinical Research, LLC, Albany, New York
  - AAIR Research Center, Rochester, New York
  - North Shore University Hospital, Valley Stream, New York
  - Appalachian Regional Medical Associates, Boone, North Carolina
  - Carolina Bone and Joint, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Hill Top Physicians Inc./Hightop Medical Research Center, Cincinnati, Ohio
  - Radiant Research, Mogadore, Ohio
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - PRO Research, Eugene, Oregon
  - School of Nursing, Portland, Oregon
  - Tri State Medical Group, Inc., Beaver, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Central Pennsylvania Clinical Research, Mechanicsburg, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Low Country Research Country, Charleston, South Carolina
  - Southern Orthopaedic Sports Medicine, Columbia, South Carolina
  - Radiant Research, Greer, Greer, South Carolina
  - Rheumatology Consultants, PLLC, Knoxville, Tennessee
  - Walter F. Chase, MD PA, Austin, Texas
  - R/D Clinical Research, Inc., Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - Radiant Research San Antonio Northeast, San Antonio, Texas
  - The University of Texas Health Science, San Antonio, Texas
  - Fatigue Consultation Center, Salt Lake City, Utah
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - Pacific Rheumatology Associates, Inc., Renton, Washington
  - Charleston Internal Medicine, Charleston, West Virginia
- France (6):
  - Rhumatologie, Amiens
  - CHU de Grenoble-Hopital Sud, Échirolles
  - Hopital Claude Huriez Service de medecine interne, Lille
  - Centre Catherine de Sienne unite d evaluation et de traitement de la douleur, Nantes
  - Hopital Hotel Dieu service de medicine interne, Paris
  - CHU Hopital de Rangueil, Toulouse
- Germany (7):
  - Gemeinschaftspraxis fur anasthesie und spezielle Schmerztherapie, Böblingen
  - Intensivmedizin der Uniklinik Koln, Cologne
  - Praxis Dr. Wiedeking, Essen
  - Praxis fur Innere Medizin und Rheumatologie, Gräfelfing
  - Gemeinschaftspraxis Schmerzzentrum, Hamburg
  - Praxisklinik Dr. Weiss, Mannheim
  - Praxis Dr. Sohn, Schwalmtal
- Azienda Ospedaliera universitaria Pisana-Ospedale Santa Chiara, Pisa, Italy
- Amphia Ziekenhuis, Breda, Netherlands
- Spain (7):
  - Hospital Santa Creu i Snt Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Instituto Ferran de Reumatologia, Barcelona
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Civil de Malaga, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
- United Kingdom (3):
  - Lever Chambers Centre for Health, Bolton
  - Kings College London, London
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Result] Spaeth M, Russell IJ, Perrot S, Alvarez-Horine S, Guinta D, Wang YG, Bennett R. Durability of Response in a 38-Week Open-Label Study of Sodium Oxybate in Patients With Fibromyalgia [ACR/ARHP abstract 2356]. Arthritis Rheum. 2010;62(suppl 10):97.
- [Derived] Spaeth M, Alegre C, Perrot S, Wang Y, Guinta DR, Alvarez-Horine S, Russell I; Sodium Oxybate Fibromyalgia Study Group. Long-term tolerability and maintenance of therapeutic response to sodium oxybate in an open-label extension study in patients with fibromyalgia. Arthritis Res Ther. 2013 Nov 11;15(6):R185. doi: 10.1186/ar4375. PMID 24286114

RESULTS

PARTICIPANT FLOW:
Groups:
- Xyrem 4.5 g to 9.0 g: Xyrem 4.5 g, 6.0 g, 7.5 g, and 9.0 g per night administered orally in two equally divided doses
Period: Overall Study
Arm/Group | Xyrem 4.5 g to 9.0 g
Started | 560
Completed | 319
Not Completed | 241
Not completed — Adverse Event | 129
Not completed — Withdrawal by Subject | 36
Not completed — Lost to Follow-up | 15
Not completed — Lack of Efficacy | 38
Not completed — Sponsor Decision | 3
Not completed — Physician Decision | 8
Not completed — Protocol Violation | 7
Not completed — Not one of the pre-specified options | 5

BASELINE CHARACTERISTICS:
Arm/Group | Xyrem 4.5 g to 9.0 g
Number analyzed (Participants) | 560
Age Continuous [Mean (Standard Deviation); unit: years] | 46.9 (10.84)
Age, Customized [Number; unit: participants]
  18 - 39 years | 144
  40 - 49 years | 181
  50 - 64 years | 212
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 510
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 34
  White | 512
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  France | 13
  United States | 465
  Spain | 35
  Netherlands | 2
  Germany | 34
  Italy | 3
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Adverse Events
Description: Number of subjects reporting adverse events.
Time Frame: Treatment Period (38 weeks)
Measure: Number; unit: Participants
Arm/Group | Xyrem 4.5 g to 9.0 g
Number analyzed (Participants) | 560
Participants | 498

ADVERSE EVENTS:
Time Frame: 38 weeks
Arm/Group | Xyrem 4.5 g to 9.0 g
Serious Adverse Events (participants affected / at risk) | 19/560
Other Adverse Events (participants affected / at risk) | 498/560
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xyrem 4.5 g to 9.0 g (N=560)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1)
Cholecystitis Chronic (Hepatobiliary disorders) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Staphylococcal Sepsis (Infections and infestations) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast Cancer in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Mental Disorder (Psychiatric disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xyrem 4.5 g to 9.0 g (N=560)
Vertigo (Ear and labyrinth disorders) | 12
Vision Blurred (Eye disorders) | 18
Nausea (Gastrointestinal disorders) | 112
Vomiting (Gastrointestinal disorders) | 52
Abdominal Pain Upper (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 24
Pyrexia (General disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 49
Oedema Peripheral (General disorders) | 13
Pain (General disorders) | 12
Nasopharyngitis (Infections and infestations) | 57
Sinusitis (Infections and infestations) | 50
Influenza (Infections and infestations) | 37
Upper Respiratory Tract Infection (Infections and infestations) | 34
Urinary Tract Infection (Infections and infestations) | 22
Bronchitis (Infections and infestations) | 18
Gastroenteritis Viral (Infections and infestations) | 16
Fall (Injury, poisoning and procedural complications) | 20
Contusion (Injury, poisoning and procedural complications) | 12
Weight Decreased (Investigations) | 21
Anorexia (Metabolism and nutrition disorders) | 16
Decreased Appetite (Metabolism and nutrition disorders) | 13
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 21
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 20
Back Pain (Musculoskeletal and connective tissue disorders) | 18
Headache (Nervous system disorders) | 106
Dizziness (Nervous system disorders) | 72
Somnolence (Nervous system disorders) | 34
Tremor (Nervous system disorders) | 20
Paraesthesia (Nervous system disorders) | 18
Migraine (Nervous system disorders) | 12
Anxiety (Psychiatric disorders) | 44
Insomnia (Psychiatric disorders) | 38
Depression (Psychiatric disorders) | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 18
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 15
Pruritus (Skin and subcutaneous tissue disorders) | 13
Hypertension (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other